CLINICAL TRIAL: NCT07034651
Title: Electron Microscopic Examination of Iris Tissue in Buphthalmos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Lotfy Fahmy, Prof, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200125
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Iris Diseases
Keywords: iris tissue, buphthalmos
MeSH Terms: conditions — Iris Diseases; Hydrophthalmos | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- isolated trabeculodysgensis (Experimental): etiology of primary congenital glaucoma
  Interventions: Procedure: Combined trabeculotomy trabeculectomy with mitomycin C

INTERVENTIONS:
Procedure: Combined trabeculotomy trabeculectomy with mitomycin C — Combined trabeculotomy trabeculectomy with mitomycin C with histopathological examination of the peripheral iris tissue specimen of all cases

SUMMARY:
To revise the etiology of the primary congenital glaucoma in some infants.

DETAILED DESCRIPTION:
Combined trabeculotomy trabeculectomy with mitomycin C was done Electron microscopic examination of the peripheral iris tissue specimen was done in all cases.

ELIGIBILITY:
Inclusion Criteria:

* infants under age of 2 years
* 1ery glaucoma

Exclusion Criteria:

* infants more than 2 years
* 2ery glaucoma
* previous glaucoma surgery

Ages: 1 Month to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
fibrovascular membrane over iris surface | 6 months
  angle closure by a fibrovascular tissue proliferation over the trabecular meshwork in the anterior chamber angle

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut univercity, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes